CLINICAL TRIAL: NCT02339272
Title: Study of Synapsis and Recombination in Male Meiosis and the Implications in Infertility
Status: Completed | Type: Observational
Sponsor: Igenomix (Industry)
Collaborators: Instituto Universitario IVI (Other)
Responsible Party: Sponsor
Other Study IDs: 070-C-027-CR
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Abnormal Spermatogenesis; Azoospermia
Keywords: meiosis; synapsis; recombination; sperm aneuploidy
MeSH Terms: conditions — Azoospermia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fixed slides with paraformaldehide, and metanol-acetic acid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NOA: Infertile males with non obstructive azoospermia
  Interventions: Other: non interventional
- OA: Post-vasectomized patients with proven fertility before vasectomy
  Interventions: Other: non interventional

INTERVENTIONS:
Other: non interventional

SUMMARY:
The aim of this study was to assess meiotic recombination in primary spermatocytes, synaptonemal complex length and the correlation with chromosomal abnormalities in testicular spermatozoa from infertile men with idiopathic non-obstructive azoospermia (NOA).

DETAILED DESCRIPTION:
During the first meiotic division in spermatogenesis there are two critical events. First, synapsis between homologous chromosomes and formation of the synaptonemal complex (SC), which regulates sister chromatid cohesion and provides the template for localization of recombination machinery proteins. Secondly, recombination between homologous chromosomes, which is essential for the correct segregation. Errors during these two processes may induce incorrect segregation of chromosomes and are a major cause of gamete aneuploidy. The aim of this study was to assess meiotic recombination in primary spermatocytes, synaptonemal complex length and the correlation with chromosomal abnormalities in testicular spermatozoa from infertile men with idiopathic non-obstructive azoospermia (NOA). Prospective cohort study to assess meiotic progression, total length of SC, frequency of recombination and sperm aneuploidy in samples obtained from testicular biopsies from NOA patients. The study group was compared with a control group from post-vasectomized (OA) patients. Immunocytogenetics with SCYP3, CREST and MLH1 antibodies for meiotic progression, SC length, and recombination. Fluorescence in situ Hybridization (FISH) for chromosomes 1, 4, 6, 13, 16, 18, 21, 22 in primary spermatocytes and chromosomes 13, 18, 21, X, Y on sperm. MicroMeasure 3.3 program was used for SC length.

ELIGIBILITY:
Inclusion Criteria:

* NOA patients undergoing ICSI with testicular sperm
* OA post-vasectomized patients undergoing ICSI with testicular sperm

Exclusion Criteria:

* Abnormal Karyotype

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Testicular biopsies from NOA patients and a control group from post-vasectomized (OA) patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Meiotic recombination | once
  Number of MLH1 foci in pachytene cells

SECONDARY OUTCOMES:
Sperm aneuploidy | once
  Percentage of sperm with aneuploidies

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Rubio, PhD, Principal Investigator — Lab Director
Locations (1):
- Igenomix, Paterna, Valencia, Spain